CLINICAL TRIAL: NCT03335735
Title: Pilot Trial Leveraging Smartphone-paired Breathalyzers and Loss- and Gain-framed Text Notifications for Reducing Drinking Driving
Brief Title: Smartphone-paired Breathalyzers and Loss- and Gain-framed Texts for Reducing Drinking and Driving
Acronym: BESAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 827345
Record Dates: First submitted 2017-10-05; First posted 2017-11-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Alcohol Drinking; Alcohol Intoxication; Alcohol Impairment; Drive; Driving Impaired; Driving Under the Influence; Behavior, Drinking
Keywords: alcohol; driving; breathalyzers; smartphone
MeSH Terms: conditions — Alcohol Drinking; Alcoholic Intoxication; Driving Under the Influence; Drinking Behavior

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant will be blinded to their random assignment into the control, loss-framed messaging, or gain-framed messaging group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Loss-Framed Text Messages (Experimental): Loss-framed text message
  Interventions: Behavioral: Loss-framed text message
- Control (No Intervention): Participants in this arm will not receive any intervention.
- Gain-Framed Messaging Group (Experimental): Gain-framed text message
  Interventions: Behavioral: Gain-Framed text message

INTERVENTIONS:
Behavioral: Loss-framed text message — Participants in the intervention group will receive loss-framed text messages related to drinking and driving on days during the week with a higher likelihood of alcohol consumption (Thursday-Saturday). Loss aversion refers to people's tendency to prefer avoiding losses to acquiring equivalent gains: it's better to not lose $5 than to find $5, so the content of the messages will be related to loss of personal freedom, loss of money, and loss of future employment opportunities due to Driving Under the Influence (DUI) convictions.
  Arms: Loss-Framed Text Messages
Behavioral: Gain-Framed text message — Participants in the intervention group will receive gain-framed text messages related to drinking and driving on days during the week with a higher likelihood of alcohol consumption (Thursday-Saturday). Gain-framed messages have been shown to have a positive effect on preventative healthcare and include content framed in a manner that the participant gains something from taking preventative action. Message content will be related to saving lives, gaining control, and making loved ones happy.
  Arms: Gain-Framed Messaging Group

SUMMARY:
This project aims to demonstrate the feasibility of a scalable behavioral intervention using smartphone-paired breathalyzers and text message aimed at reducing drinking and driving among individuals who report heavy drinking. All participants receive a smartphone breathalyzer to provide feedback on their estimated blood alcohol level. The intervention compares loss- and gain-framed messages that make the consequences of drinking and driving more salient to standard messages not to drink and drive.

DETAILED DESCRIPTION:
The overall objective of this project is to leverage smartphone-paired breathalyzers to implement cost-effective and scalable behavioral interventions to reduce risky drinking behaviors such as drinking and driving. Prospect theory proposes that messages framed in different ways can elicit different responses from individuals. Loss aversion refers to people's tendency to prefer avoiding losses to acquiring equivalent gains: it's better to not lose $5 than to find $5. People are more motivated to avoid losing something than they are to win something. Studies have found that delivering messaging framed as a loss are also effective in motivating certain behaviors. On the other hand, gain-framed messages have been shown to have a positive effect on preventative healthcare. By using automated remote monitoring, innovative loss aversion and gain-framed messaging strategies incorporating insights from behavioral economics could be more easily implemented by delivering effective messaging prior to a risky behavior taking place. The investigators hope that the use of loss aversive and/or gain-framed messaging will lead to individuals improving planning behavior around drinking, especially in regards to drinking and driving. The objective of this project is to demonstrate the feasibility of a scalable intervention using loss- gain-framed messaging to reduce drinking and driving, compare the effectiveness of each type of messaging, and to increase the use of Blood Alcohol Content (BAC) monitors as a way to plan safer strategies when drinking. The investigators' long-term objective is to secure federal funding for research that leverages insights from behavioral economics supported by smartphone technology to reduce risky drinking.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 21-39
* Reports an average of one heavy drinking day (men more than five drinks, women more than four drinks) per week over the preceding 8 weeks
* Has a valid photo identification (ID)
* Are willing and able to use an Uber or Lyft or septa as transportation home
* Drives four or more trips per week
* Owns an Apple iPhone or Android smartphone

Exclusion Criteria:

* Desire for alcohol treatment now or have received alcohol treatment within the past 6 months
* Alcohol use disorder rated as severe per DSM-V criteria
* Non-English-speaking
* Women who are pregnant
* Individuals who should not consume alcohol due to a medical condition such as liver disease, cancer, and seizure disorders. Participants will be asked to answer yes if they have any disorder that their doctor has suggested that they should not drink alcohol. If they are unsure or say I don't know the investigators will ask them to speak with their doctor prior to participation.

Ages: 21 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the change in proportion of breathalyzer measurements submitted with self-reported drinking episodes across groups. | baseline up to 8 weeks

SECONDARY OUTCOMES:
Change in frequency of BACtrack monitoring within intervention group from baseline | baseline up to 8 weeks
Drinking and driving episodes in which their BAC via self-report or BAC measure is expected to be positive | baseline up to 8 weeks
  To be assessed using a driving monitoring app passively running on participants' phones throughout the trial
Changes in accuracy of BAC guess vs actual BAC measure with continued use (Does a participant become more accurate overtime in predicting what their BAC will be prior to measuring) | baseline up to 8 weeks
  Participants are able to guess their BAC within the app before collecting the measurement. We will examine the changes in the accuracy of their guesses over time

CONTACTS AND LOCATIONS:
Overall Officials: Kit Delgado, MD, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers. In fact, there will be an NIH Certificate of Confidentiality protecting participants' data.

REFERENCES:
- [Background] White A, Hingson R. The burden of alcohol use: excessive alcohol consumption and related consequences among college students. Alcohol Res. 2013;35(2):201-18. doi: 10.35946/arcr.v35.2.11. PMID 24881329
- [Background] Sloan FA, Eldred LM, Xu Y. The behavioral economics of drunk driving. J Health Econ. 2014 May;35:64-81. doi: 10.1016/j.jhealeco.2014.01.005. Epub 2014 Feb 11. PMID 24603444
- [Background] Naimi TS, Brewer RD, Mokdad A, Denny C, Serdula MK, Marks JS. Binge drinking among US adults. JAMA. 2003 Jan 1;289(1):70-5. doi: 10.1001/jama.289.1.70. PMID 12503979
- [Background] Matjasko JL, Cawley JH, Baker-Goering MM, Yokum DV. Applying Behavioral Economics to Public Health Policy: Illustrative Examples and Promising Directions. Am J Prev Med. 2016 May;50(5 Suppl 1):S13-S19. doi: 10.1016/j.amepre.2016.02.007. PMID 27102853
- [Background] Schneider TR, Salovey P, Apanovitch AM, Pizarro J, McCarthy D, Zullo J, Rothman AJ. The effects of message framing and ethnic targeting on mammography use among low-income women. Health Psychol. 2001 Jul;20(4):256-66. doi: 10.1037//0278-6133.20.4.256. PMID 11515737
- [Background] Toll BA, O'Malley SS, Katulak NA, Wu R, Dubin JA, Latimer A, Meandzija B, George TP, Jatlow P, Cooney JL, Salovey P. Comparing gain- and loss-framed messages for smoking cessation with sustained-release bupropion: a randomized controlled trial. Psychol Addict Behav. 2007 Dec;21(4):534-44. doi: 10.1037/0893-164X.21.4.534. PMID 18072836
- [Background] List JA, Samek AS. The behavioralist as nutritionist: leveraging behavioral economics to improve child food choice and consumption. J Health Econ. 2015 Jan;39:135-46. doi: 10.1016/j.jhealeco.2014.11.002. Epub 2014 Nov 21. PMID 25530206
- [Background] MacKillop J, Amlung MT, Few LR, Ray LA, Sweet LH, Munafo MR. Delayed reward discounting and addictive behavior: a meta-analysis. Psychopharmacology (Berl). 2011 Aug;216(3):305-21. doi: 10.1007/s00213-011-2229-0. Epub 2011 Mar 4. PMID 21373791
- [Background] Petry NM, Martin B, Cooney JL, Kranzler HR. Give them prizes, and they will come: contingency management for treatment of alcohol dependence. J Consult Clin Psychol. 2000 Apr;68(2):250-7. doi: 10.1037//0022-006x.68.2.250. PMID 10780125
- [Background] Loewenstein G, Brennan T, Volpp KG. Asymmetric paternalism to improve health behaviors. JAMA. 2007 Nov 28;298(20):2415-7. doi: 10.1001/jama.298.20.2415. No abstract available. PMID 18042920
- [Background] Patel MS, Asch DA, Volpp KG. Wearable devices as facilitators, not drivers, of health behavior change. JAMA. 2015 Feb 3;313(5):459-60. doi: 10.1001/jama.2014.14781. No abstract available. PMID 25569175
- [Background] Sobell LC, Brown J, Leo GI, Sobell MB. The reliability of the Alcohol Timeline Followback when administered by telephone and by computer. Drug Alcohol Depend. 1996 Sep;42(1):49-54. doi: 10.1016/0376-8716(96)01263-x. PMID 8889403
- [Background] Case MA, Burwick HA, Volpp KG, Patel MS. Accuracy of smartphone applications and wearable devices for tracking physical activity data. JAMA. 2015 Feb 10;313(6):625-6. doi: 10.1001/jama.2014.17841. No abstract available. PMID 25668268
- [Background] South EC, Kondo MC, Cheney RA, Branas CC. Neighborhood blight, stress, and health: a walking trial of urban greening and ambulatory heart rate. Am J Public Health. 2015 May;105(5):909-13. doi: 10.2105/AJPH.2014.302526. Epub 2015 Mar 19. PMID 25790382
- [Background] Byrnes HF, Miller BA, Wiebe DJ, Morrison CN, Remer LG, Wiehe SE. Tracking Adolescents With Global Positioning System-Enabled Cell Phones to Study Contextual Exposures and Alcohol and Marijuana Use: A Pilot Study. J Adolesc Health. 2015 Aug;57(2):245-7. doi: 10.1016/j.jadohealth.2015.04.013. PMID 26206448
- [Background] Patel MS, Asch DA, Rosin R, Small DS, Bellamy SL, Heuer J, Sproat S, Hyson C, Haff N, Lee SM, Wesby L, Hoffer K, Shuttleworth D, Taylor DH, Hilbert V, Zhu J, Yang L, Wang X, Volpp KG. Framing Financial Incentives to Increase Physical Activity Among Overweight and Obese Adults: A Randomized, Controlled Trial. Ann Intern Med. 2016 Mar 15;164(6):385-94. doi: 10.7326/M15-1635. Epub 2016 Feb 16. PMID 26881417
- See also: BacTrack Mobile Pro breathalyzer device — http://www.bactrack.com/products/bactrack-mobile-breathalyzer?gclid=Cj0KEQiAzO6zBRC25Ju1idGJiZkBEiQAP3Sf6MVZKaULJEmXCJnBgqXvqrzfuiYe3hpIEsgMir1_QXUaAl_o8P8HAQ
- See also: Centers for Disease Control and Prevention. BRFSS Prevalence & Trends Data.; 2015 — http://www.cdc.gov/brfss/brfssprevalence

DOCUMENTS (2):
  • Study Protocol (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT03335735/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT03335735/SAP_001.pdf